CLINICAL TRIAL: NCT05003063
Title: Effects of Acetylcholine and Attention on Visual Spatial Representations in the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018-10-11532
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Visual Perception; Attention; Information Processing; Cholinergic System
Keywords: Attention; Visual Perception; Cholinergic system

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Donepezil (Active Comparator): 5mg Donepezil will be administered in pill form.
  Interventions: Drug: Donepzil
- Placebo (Placebo Comparator): 5mg placebo will be administered in pill form.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Donepzil — Test
  Arms: Donepezil
Drug: Placebo oral tablet — Test
  Arms: Placebo

SUMMARY:
This study in, healthy human subjects using fMRI and MRS (magnetic resonance spectroscopy) characterizes, how attention and acetylcholine affect visual perception and the brain's representation of the visual environment. Levels of acetylcholine in the cerebral cortex will be enhanced by administration of donepezil, an inhibitor of acetylcholinesterase. Half the subjects will receive donepezil and other half will receive placebo.

DETAILED DESCRIPTION:
The long-term objective of this project is to characterize how attention and acetylcholine affect visual perception and the brain's representation of the visual environment. Acetylcholine is a naturally occurring neurotransmitter, and acetylcholine release is elevated during periods of sustained attention. Both acetylcholine and attention enhance aspects of visual perception, but the underlying brain mechanisms are poorly understood. The proposed work will address these questions in healthy human subjects by using functional magnetic resonance imaging (fMRI) and MRS (magnetic resonance spectroscopy) to measure the brain's responses to visual stimuli. Our previous studies have shown that increasing levels of acetylcholine in the brain enhances the spatial resolution of the brain's representation of the visual environment. The proposed research will document exactly which brain areas mediate this effect of acetylcholine and will also characterize the effects of attention on these measures of spatial resolution in the brain.

The technique of fMRI (functional magnetic resonance imaging) and MRS (magnetic resonance spectroscopy), both subtypes of MRI, will be employed to measure brain activity in different brain areas while subjects are performing a visual attention task. Levels of acetylcholine in the cerebral cortex will be enhanced by administration of donepezil, an inhibitor of acetylcholinesterase, the enzyme that metabolizes acetylcholine. Moreover, the technique of MRS will be employed to locally quantify the levels of acetylcholine in different brain areas.

In addition to providing information about how attention is represented in the brain and how it affects processing of visual stimuli, the present experiments should also shed light on the function of the cholinergic projection from the basal forebrain to the cerebral cortex. As this projection is thought to be selectively impaired in Alzheimer's disease, knowledge concerning its function in the healthy brain may be useful for understanding the etiology of this disease and for development of appropriate therapies.

BEHAVIORAL PHARMACOLOGY:

Sessions:

Subjects will perform 6 behavioral sessions over several days outside the scanner, split into two experimental parts. There will be 2 baseline sessions without donepezil/placebo and 4 testing sessions with donepezil/placebo. Each behavioral (outside the scanner) session will last 1-2 hours. During the testing session, subjects will be given one pill of (2.5 or 5 or 10mg) donepezil or placebo per session. The choice of the pill will be determined by the flip of a coin. The drug dosage (2.5 or 5 or 10mg) will be determined so as to ensure that there are equal number of participants per drug dosage. The pill (drug or placebo) not selected for the first experimental session in a pair will be administered during the second experimental session.

Task:

A typical cognitive task will involve presentation of images or words on a computer monitor or sounds through headphones. The subjects are asked to respond to certain stimuli by pressing a button. All stimuli are presented at a comfortable level. The cognitive task performed during the behavioral is an object-tracking/target detection paradigm in which subjects indicate whether a target is presented or not on each experimental trial. The target, when it is presented, is a visual stimulus at the threshold of detectability. On some trials, subjects will receive cues indicating target location and/or features that will facilitate target detection. Subjects will be asked to report by pressing a button on a response box. Subjects will receive breaks every 5-10 minutes or more frequently if they desire.

MRI AND PHARMACOLOGY:

Sessions:

For experiments involving MRI, there will be a total of 6 sessions across several days, split into two experimental parts. There will be two baseline MRI session without donepezil/placebo and 4 testing sessions (two donepezil, two placebo). Subjects will be given one pill of (2.5 or 5 or 10mg) donepezil or placebo per session. The choice of the pill will be determined by the flip of a coin. The pill not selected for the first experimental part will be administered during the second experimental part.

For MRI experiments, the experimenter will escort the subject to the Brain Imaging Center in Li Ka Shing about 2.5 hours after pill administration, and fMRI measurements will begin approximately 3 hours after pill administration. The MRI sessions typically take 1-2.5 hours, and the subject is given frequent breaks. The subject may stop the experiment at any time. Subjects undergoing MRI scanning will be asked to lie on their back in the MRI scanner. Before being scanned, a MRI imaging coil made of plastic will be placed around the subject's head. The subject will not come into contact with the coil during the experiment. Foam pads will be placed around the subject's head to limit head movement during the study.

Task:

A typical cognitive task will involve presentation of images or words on a computer monitor or sounds through headphones. The subjects are asked to respond to certain stimuli by pressing a button. All stimuli are presented at a comfortable level. The cognitive task performed during the behavioral is an object-tracking/target detection paradigm in which subjects indicate whether a target is presented or not on each experimental trial. The target, when it is presented, is a visual stimulus at the threshold of detectability. On some trials, subjects will receive cues indicating target location and/or features that will facilitate target detection. Subjects will be asked to report by pressing a button on a response box. Subjects will receive breaks every 5-10 minutes or more frequently if they desire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult individuals

Exclusion Criteria:

* Pregnancy
* Asthma/lung problems
* Certain medications, seizure
* Failure to complete Donepezil (Aricept) Contraindications Screening Sheet
* Previous long term exposure to nicotine/tobacco products, individuals with pacemakers, cosmetics, or certain metallic implants in their bodies will be excluded from experiments involving MRI recording.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Population receptive field (pRF) size | Starting 3 hours after pill administration. 1 functional scan every 4 minutes for one hour.
  measuring pRF size changes due to donepezil intervention

SECONDARY OUTCOMES:
Population receptive field (pRF) eccentricity | Starting 3 hours after pill administration. 1 functional scan every 4 minutes for one hour.
  measuring pRF eccentricity changes due to donepezil intervention
Response amplitude | Starting 3 hours after pill administration. 1 functional scan every 4 minutes for one hour.
  measuring Response amplitude changes due to donepezil intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided